CLINICAL TRIAL: NCT05707026
Title: Comparative Effects of Cross Fiber Fascial Manipulation and Stretching Techniques on Glenohumeral Internal Rotation Deficit in Overhead Throwing Athletes
Brief Title: Cross Fiber Fascial Manipulation and Stretching Techniques in Overhead Throwing Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0408
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Overhead Throwing Athletes; Tennis Players, Bowlers, Volleyball Players

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cross fiber fascial manipulation (Experimental): The group A received three sessions of fascial manipulation in two weeks. FM applied to densified Centre of Coordination (CC) points located on the myofascial sequences for 5 to 8 minutes at each CC point
  Interventions: Other: cross fiber fascial manipulation
- stretching techniques (Experimental): Group B received three sessions of sleeper and cross body adduction stretches. Group B received three sessions of sleeper stretch in a side lying position in 90o abduction, elbow at 90o flexion and then performing shoulder IR and cross-body adduction stretch was done in sitting position. Three sets of the each stretch position were held for 30 seconds with a 1 minute break between sets
  Interventions: Other: stretching techniques(sleeper stretch and cross body adduction stretch)

INTERVENTIONS:
Other: cross fiber fascial manipulation — The group A received three sessions of fascial manipulation in two weeks. FM applied for 5 to 8 minutes at each point.
  Arms: cross fiber fascial manipulation
Other: stretching techniques(sleeper stretch and cross body adduction stretch) — Group B received three sessions of sleeper and cross body adduction stretches. Group B received three sessions of sleeper stretch in a side lying position in 90o abduction, elbow at 90o flexion and then performing shoulder IR and cross-body adduction stretch was done in sitting position. Three sets of the each stretch position were held for 30 seconds with a 1 minute break between sets.
  Arms: stretching techniques

SUMMARY:
Athletic training and sports participation is to enhance athletic performance. Performance is however multifactorial i.e., depending upon several parameters including warm-up practice, training regimes and other interventions. Stretching techniques that focus on increasing posterior shoulder soft tissue flexibility are commonly incorporated into prevention and treatment programs for the overhead athletes. GIRD is usually managed by stretching and soft tissue release of posterior shoulder capsule. Fascial manipulation is a manual therapy technique used in the management of musculoskeletal disorders. This study aims to evaluate the comparative effects of cross fiber fascial manipulation with stretching techniques in overhead throwing athletes

DETAILED DESCRIPTION:
This was a randomized clinical trial that was conducted at Pakistan sports board and Coaching center, Lahore. Non probability convenient sampling technique was used to collect the data as per inclusion criteria. 40 Participants of this study were randomly allocated into 2 Groups. 20 participants in each group. The group A received three sessions of fascial manipulation for two weeks. Group B received three sessions of sleeper stretch in a side lying position in 90o abduction, elbow at 90o flexion and then performed shoulder IR and cross-body adduction stretch in sitting position. Three sets of the each stretch positions were held for 30 seconds with a 1 minute break between sets. A universal goniometer was used to measure internal rotation, external rotation, horizontal abduction, ROWE score to assess function, pain, stability and motion, Numeric pain rating scale (NPRS) was used to assess pain. The data was analyzed via SPSS version 22.

ELIGIBILITY:
Inclusion Criteria:

* Active male and female athletes were included.

  * Age group was (18-40) .
  * Overhead throwing athletes(tennis, volleyball, bowlers) were included in this study)
  * Screening tests were taken to identify subjects with GIRD. GIRD was defined as more than 20o decrease in IR at 90o abduction in the dominant side compared to non-dominant side .
  * Subjects who rated shoulder pain 5 or more in NPRS/symptomatic with GIRD were recruited

Exclusion Criteria :

* Any deformity
* Any radiculopathy
* Shoulder traumatic injuries( dislocation, subluxation, fracture)
* Systemic illness
* Subacromial impingement signs

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Goniometer | 2 weeks
  A universal goniometer was used to assess internal rotation, external rotation and horizontal adduction
numeric pain rating scale | 2 weeks
  NPRS for pain assessment in overhead athletes reporting pain with GIRD, it is a subjective measure in which individual rate their pain on an 11-point numerical scale. The scale is composed of 0 (no pain at all) to 10( worst pain
ROWE score composite | 2 weeks
  ROWE score for shoulder functional assessment(50), stability(30), pain(10) and motion(10). Total score is 100 thus 90-100=excellent ,70-89=good , 40-69=fair , less than 40 points=poor

CONTACTS AND LOCATIONS:
Overall Officials: aqsa nawaz, MS SPORTS pt, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No